CLINICAL TRIAL: NCT01472484
Title: A Stable Iron Isotope Study to Investigate the Impact of Phytic Acid and Polyphenols on Iron Absorption From Beans in Humans
Brief Title: Impact of Bean Polyphenols and Phytic Acid on Iron Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: lpa_586/8X87
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Blood Iron Isotope Enrichment
Keywords: beans; lpa mutant; polyphenols; phytic acid; stable iron isotopes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- lpa with high polyphenol (Experimental)
  Interventions: Other: 586/8x87 brown
- lpa with low polyphenol (Experimental)
  Interventions: Other: 586/8x87 white
- control bean with low polyphenol (Experimental)
  Interventions: Other: 586/8
- control bean with high polyphenol (Experimental)
  Interventions: Other: BAT 881

INTERVENTIONS:
Other: 586/8x87 white — 2 x 50 g
  Arms: lpa with low polyphenol
Other: 586/8x87 brown — 2 x 50 g
  Arms: lpa with high polyphenol
Other: BAT 881 — 2 x 50 g
  Arms: control bean with high polyphenol
Other: 586/8 — 2 x 50 g
  Arms: control bean with low polyphenol

SUMMARY:
Recently isolated low PA varieties (lpa) in wheat, rice, maize, barley and beans might have the potential to alleviate iron bioavailability problems associated with PA. These plants have normal phosphate levels, but reduced PA phosphate due to various modifications of the biosynthetic pathway of PA. So far lpa crops are in an early stage of development, most of them exhibiting reduced yield and seed germination. However, the lpa bean isolated by Campion and co-workers 2009 by chemical mutagenesis exhibited only 10 % of the native bean PA concentration without any defects in terms of growth and yield.

Crossing the lpa variety with bean varieties low in PP and high in iron might lead to the development of a variety which has the potential to improve the iron status of bean consuming populations.

The following study will evaluate the relative impact of PA and PP on iron absorption from beans by comparing iron absorption from four different bean varieties. Iron absorption from a bean with normal PA concentration and high PP concentration will be compared to iron absorption from a bean with normal PA and low PP concentration as well as to two lpa varieties, one with high and one with low PP concentration.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-lactating women
* Between 18 and 40 years
* Below 65kg

Exclusion Criteria:

* Metabolic, chronic and gastro-intestinal disease
* Long-term medication
* Blood donation within 6 month before the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Shift in iron isotopic composition in blood after consumption of different bean varieties | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hurrell, Prof. Dr., Principal Investigator — ETH Zürich
Locations (1):
- ETH, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Petry N, Egli I, Campion B, Nielsen E, Hurrell R. Genetic reduction of phytate in common bean (Phaseolus vulgaris L.) seeds increases iron absorption in young women. J Nutr. 2013 Aug;143(8):1219-24. doi: 10.3945/jn.113.175067. Epub 2013 Jun 19. PMID 23784069